CLINICAL TRIAL: NCT02466503
Title: A Single-Dose, Randomized, Open-Label, Crossover, Pivotal, Comparative Bioavailability Study of Synflutide HFA 250/25 Inhaler and SeretideTM 250 EvohalerTM in Healthy Volunteers With Charcoal Block
Brief Title: Bioequivalence Study of Synflutide HFA Inhaler and Seretide Evohaler in Healthy Volunteers With Charcoal Block
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCPE14015M1
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synflutide HFA MDI, 250/25 mcg/dose (Experimental): Synflutide HFA MDI(Fluticasone propionate/ Salmeterol, 250/25mcg), Single dose, 4 puffs
  Interventions: Drug: Fluticasone propionate; Drug: Salmeterol (as xinafoate)
- SeretideTM EvohalerTM, 250/25 mcg/dose (Active Comparator): SeretideTM EvohalerTM (Fluticasone propionate/ Salmeterol, 250/25mcg), Single dose, 4 puffs
  Interventions: Drug: Fluticasone propionate; Drug: Salmeterol (as xinafoate)

INTERVENTIONS:
Drug: Fluticasone propionate — Inhaled corticosteroid, pMDI
  Other Names: Flovent; Flixotide
Drug: Salmeterol (as xinafoate) — Beta-agonist, LABA, pMDI
  Other Names: Serevent

SUMMARY:
The objective of this pivotal study is to evaluate the relative bioavailability of Synflutide HFA 250/25 Inhaler and SeretideTM 250 EvohalerTM in healthy volunteers with charcoal block.

DETAILED DESCRIPTION:
A pivotal, single-dose, randomized, open-label, two-period, two-sequence, two-treatment, crossover, comparative bioavailability study for test drug Synflutide HFA 250/25 Inhaler and reference drug SeretideTM 250 EvohalerTM in healthy volunteers with charcoal block. Fifty healthy, male and female volunteers, 20-65 years of age, with a body mass index (BMI) within 18.0-30.0 kg/m2, inclusive, will be enrolled. A single dose of 4 puffs (eq. to fluticasone propionate 1000μg+salmeterol 100μg from valve) in each study period. Plasma samples will be assayed for fluticasone propionate and salmeterol using a validated analytical method according to the principles of Good Laboratory Practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, aged 20-65, inclusive.
* BMI that is within 18.0-30.0 kg/m², inclusive.
* Healthy or Non Clinical Significant, according to the medical history, ECG, Chest X-ray and physical examination as determined by the Principal Investigator/Sub-Investigator.
* Systolic blood pressure between 90-139 mmHg, inclusive, and diastolic blood pressure between 50-90 mmHg, inclusive, and pulse rate between 50-100 bpm, inclusive and temperature between 35.0-37.4℃.
* Clinical laboratory values within PPC's acceptable range according to PPC SOP VI-006.
* Ability to comprehend and be informed of the nature of the study, as assessed by PPC staff. Capable of giving written informed consent prior to receiving any study medication. Must be able to communicate effectively with clinic staff.
* Ability to fast for at least 14 hours and to consume standard meals.
* Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
* Agree not to have a tattoo or body piercing until the end of the study.
* Female subjects must fulfill at least one of the following:

  * Be surgically sterile for a minimum of 6 months;
  * Post-menopausal for a minimum of 1 year;
  * Agree to avoid pregnancy and use medically acceptable method of contraception from at least 30 days prior to the study until 30 days after the study has ended (last study procedure).

Exclusion Criteria:

* Known history or presence of any clinically significant hepatic (e.g. active liver disease, hepatic impairment), renal/genitourinary (e.g. renal impairment), gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine (e.g. hypothyroidism), immunological, musculoskeletal (e.g. myopathy, rhabdomyolysis), neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the Principal Investigator/Sub-Investigator.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first drug administration, as determined by the Principal Investigator/Sub-Investigator.
* Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the Principal Investigator/Sub-Investigator.
* Presence of any significant physical or organ abnormality as determined by the Principal Investigator/Sub-Investigator.
* A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine, tetrahydrocannabinol), breath alcohol test. Positive pregnancy test for female subjects.
* Known history or presence of:

  * Alcohol abuse or dependence within one year prior to first drug administration;
  * Drug abuse or dependence;
  * Hypersensitivity or idiosyncratic reaction to fluticasone propionate, salmeterol xinafoate, its excipients, and/or related substances;
  * Food allergies and/or presence of any dietary restrictions;
  * Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
* Intolerance to and/or difficulty with blood sampling through venipuncture.
* Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets etc.
* Individuals who have donated, in the days prior to first drug administration:

  * Less than 250 mL of blood in the previous 60 days
  * 300 mL or more in the previous 90 days
* Donation of plasma by plasmapheresis within 7 days prior to first drug administration.
* Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first drug administration.
* Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing and containing grapefruit and/or pomelo within 10 days prior to first drug administration.
* Use of any prescription medication or investigational medication within 30 days prior to first drug administration.
* Use of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 30 days prior to first drug administration (except for spermicidal/barrier contraceptive products).
* Females taking oral or transdermal hormonal contraceptives within 30 days prior to first drug administration.
* Females having used implanted, injected, intravaginal, or intrauterine hormonal contraceptive within 6 months prior to first drug administration.
* Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by Principal Investigator/Sub-Investigator.
* Known history of smoking or using tobacco products, nicotine products (patches, gum etc.) within 6 months prior to first drug administration.
* Pregnant/lactating women.
* Subjects will be given training to ensure that subjects are able to correctly use the investigational products in screening. The subjects who are unable to operate the investigational products proficiently will not be included in this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Pre-dose and at 0.08, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after dosing
Maximum plasma concentration (Cmax) | Pre-dose and at 0.08, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after dosing

SECONDARY OUTCOMES:
Time to reach Maximum plasma concentration (Tmax) | Pre-dose and at 0.08, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 and 24 hours after dosing
blood pressure [BP] | pre-dose and 0.5, 2 and 24 hours after dosing
pulse rate [PR] | pre-dose and 0.5, 2 and 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: W K Chang, M.D, Principal Investigator — Clinical Pharmacology Unit of Mackay Memorial Hospital Tamshui Branch
Locations (1):
- Clinical Pharmacology Unit of Mackay Memorial Hospital Tamshui Branch, New Taipei City, Taiwan